CLINICAL TRIAL: NCT05107232
Title: OSV-IRM - Volunteer MRI Sequence Optimization
Acronym: OSV-IRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC21_8958_OSV-IRM
Record Dates: First submitted 2021-10-06; First posted 2021-11-04 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): Patients and Healthy volunteers included will have an MRI
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI

SUMMARY:
Optimization of magnetic resonance imaging (MRI) protocols on healthy volunteers and voluntary patients.

In MRI, a large number of technical parameters (sequence, parameters in sequence, antenna, reconstruction method, etc.) can be changed to optimize the diagnostic quality of the exam. Some optimizations can be performed on participants healthy volunteers, others need to be carried out on images pathological and acquired in voluntary patients.

DETAILED DESCRIPTION:
An inclusion visit is planned to verify the criteria for selection, then an imaging visit to perform the MRI examination.

The imaging visit can take place at the end of the inclusion visit and until the following 15 days. For healthy volunteers, the visits are organized according to their availability. For patients, on the other hand, participation in the research will depend on the programming of the MRI within the framework care.

This is a single-center prospective study carried out at two sites in the Rennes University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Criteria common to all participants:

  * Minor or major subject
  * Affiliated, himself or through his parents if he is a minor, to a a social security scheme
  * Having given their free, informed and written consent, and/or which the free, informed and written consent of the holder(s) parental authority has been obtained for minors

Specific criteria for healthy volunteers:

o No medical or surgical history related to the anatomical area(s) scanned

Specific criteria for voluntary patients:

o Indication for an MRI exam as part of its management

Exclusion Criteria:

* - Contraindication to an MRI (pacemaker or pacemaker, neurostimulator, intra-orbital metal body, vascular clip ferromagnetic)
* Pregnancy
* Legal protection measure for adults in progress (safeguard of justice, guardianship, curatorship) or subject deprived of liberty

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quality of MRI signal | 15 days
  The quality of the images, maps or signals collected will be compared to standard acquisitions. This evaluation will be done by statistical comparison of visual qualitative criteria by expert radiologists or on quantitative criteria drawn from analyzes computing data obtained by processing experts images (signal-to-noise ratio, contrast-to-noise ratio, blur level, mutual information, co-location of regions highlighted by different techniques, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe FERRE, Pr, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided